CLINICAL TRIAL: NCT00996736
Title: Mycotic Ulcer Treatment Trial
Brief Title: Mycotic Ulcer Treatment Trial I
Acronym: MUTT I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Aravind Eye Hospitals, India (Other); Dartmouth-Hitchcock Medical Center (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Thomas M. Lietman, Professor in Residence, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H9332-33965-02; U10EY018573-01A1 (NIH)
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Corneal Ulcer; Eye Infections, Fungal
Keywords: Fungal Infections; Eye Disease; Fungal Keratitis; Visual Acuity
MeSH Terms: conditions — Corneal Ulcer; Eye Infections, Fungal; Mycoses; Eye Diseases | interventions — Natamycin; Voriconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Natamycin (Active Comparator)
  Interventions: Drug: Natamycin
- Topical Voriconazole (Experimental)
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Natamycin — 5% natamycin plus 0.02% preservative, one drop to the affected eye every one hour while awake for 1 week, then every 2 hours while awake until 3 weeks after enrollment.
  Arms: Topical Natamycin
Drug: Voriconazole — 1% voriconazole plus 0.01% preservative, 1 drop applied to the affected eye every one hour while awake for 1 week, then every 2 hours while awake until three weeks after enrollment.
  Arms: Topical Voriconazole

SUMMARY:
The purpose of this study is to determine if natamycin or voriconazole results in better visual outcomes in fungal corneal ulcers, especially visual acuity.

DETAILED DESCRIPTION:
Fungal corneal ulcers tend to have very poor outcomes with commonly used treatments. There has only been a single randomized trial of anti-fungal therapy for mycotic keratitis, and no new ocular anti-fungal medications have been approved by the FDA since the 1960s. The triazole voriconazole has recently become the treatment of choice for systemic fungal infections such as pulmonary aspergillosis. The use of topical ophthalmic preparations of voriconazole has been described in numerous case reports, however there has been no systematic attempt to determine whether it is more or less clinically effective than natamycin. Additionally, there have been many case reports of the use of oral voriconazole in the treatment of fungal corneal ulcers, however there has been no systematic attempt to determine if it improves outcomes in severe ulcers.

This study is a randomized, double-masked, placebo-controlled trial to determine if the use natamycin or voriconazole results in better outcomes for fungal corneal ulcers. 368 fungal corneal ulcers with baseline visual acuity between 6/12 (20/40, logMAR 0.3) and 6/120 (20/400, logMAR 1.3) presenting to the Aravind Eye Hospitals and the UCSF Proctor Foundation will be randomized to receive either topical natamycin or topical voriconazole. The primary outcome is best spectacle-corrected logMAR visual acuity three months after enrollment, using best spectacle-corrected enrollment visual acuity as a co-variate.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a corneal ulcer at presentation
* Evidence of filamentous fungus on smear (KOH wet mount, Giemsa, or Gram stain)
* Visual acuity between 6/12 (20/40, logMAR 0.3) and 6/120 (20/400, logMAR 1.3)
* The patient must be able to verbalize a basic understanding of the study after it is explained to the patient, as determined by physician examiner. This understanding must include a commitment to return for follow-up visits.
* Willingness to be treated as an inpatient or to be treated as an outpatient and return every 3 days +/- 1 day until re-epithelialization and every week to receive fresh medication for 3 weeks
* Appropriate consent

Exclusion Criteria:

* Impending perforation
* Evidence of bacteria on Gram stain at the time of enrollment
* Evidence of acanthamoeba by stain
* Evidence of herpetic keratitis by history or exam
* Corneal scar not easily distinguishable from current ulcer
* Age less than 16 years (before 16th birthday)
* Bilateral ulcers
* Previous penetrating keratoplasty in the affected eye
* Pregnancy (by history or urine test) or breast feeding (by history)
* Acuity worse than 6/60 (2/200) in the fellow eye (note that any acuity, uncorrected, corrected, pinhole, or BSCVA 6/60 or better qualifies for enrollment)
* Acuity worse than 6/120 (20/400) or better than 6/12 (20/40) in the study eye (note that any acuity, uncorrected, corrected, pinhole, or BSCVA can be used for enrollment)
* Known allergy to study medications (antifungal or preservative)
* No light perception in the affected eye
* Not willing to participate

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NV Prajna, DNB, FRC Ophth, Principal Investigator — Aravind Eye Hospitals; Nisha Acharya, MD, MS, Principal Investigator — Proctor Foundation, UCSF; Tom Lietman, MD, Principal Investigator — Proctor Foundation, UCSF
Locations (3):
- Proctor Foundation, UCSF, San Francisco, California, United States
- India (2):
  - Aravind Eye Hospitals, Madurai, Tamil Nadu
  - Aravind Eye Hospital, Pondicherry, Tamil Nadu

REFERENCES:
- [Background] Prajna NV, Krishnan T, Mascarenhas J, Rajaraman R, Prajna L, Srinivasan M, Raghavan A, Oldenburg CE, Ray KJ, Zegans ME, McLeod SD, Porco TC, Acharya NR, Lietman TM; Mycotic Ulcer Treatment Trial Group. The mycotic ulcer treatment trial: a randomized trial comparing natamycin vs voriconazole. JAMA Ophthalmol. 2013 Apr;131(4):422-9. doi: 10.1001/jamaophthalmol.2013.1497. PMID 23710492
- [Derived] Prajna NV, Lalitha P, Krishnan T, Rajaraman R, Radnakrishnan N, Srinivasan M, Devi L, Das M, Liu Z, Zegans ME, Acharya NR, Porco TC, Lietman TM, Rose-Nussbaumer J. Patterns of Antifungal Resistance in Adult Patients With Fungal Keratitis in South India: A Post Hoc Analysis of 3 Randomized Clinical Trials. JAMA Ophthalmol. 2022 Feb 1;140(2):179-184. doi: 10.1001/jamaophthalmol.2021.5765. PMID 35024776
- [Derived] Prajna NV, Krishnan T, Rajaraman R, Patel S, Shah R, Srinivasan M, Das M, Ray KJ, Oldenburg CE, McLeod SD, Zegans ME, Acharya NR, Lietman TM, Rose-Nussbaumer J; Mycotic Ulcer Treatment Trial Group. Predictors of Corneal Perforation or Need for Therapeutic Keratoplasty in Severe Fungal Keratitis: A Secondary Analysis of the Mycotic Ulcer Treatment Trial II. JAMA Ophthalmol. 2017 Sep 1;135(9):987-991. doi: 10.1001/jamaophthalmol.2017.2914. PMID 28817744
- [Derived] Prajna NV, Krishnan T, Rajaraman R, Patel S, Shah R, Srinivasan M, Devi L, Das M, Ray KJ, O'Brien KS, Oldenburg CE, McLeod SD, Zegans ME, Acharya NR, Lietman TM, Rose-Nussbaumer J; Mycotic Ulcer Treatment Trial Group. Adjunctive Oral Voriconazole Treatment of Fusarium Keratitis: A Secondary Analysis From the Mycotic Ulcer Treatment Trial II. JAMA Ophthalmol. 2017 Jun 1;135(6):520-525. doi: 10.1001/jamaophthalmol.2017.0616. PMID 28426856
- [Derived] Prajna NV, Krishnan T, Rajaraman R, Patel S, Srinivasan M, Das M, Ray KJ, O'Brien KS, Oldenburg CE, McLeod SD, Zegans ME, Porco TC, Acharya NR, Lietman TM, Rose-Nussbaumer J; Mycotic Ulcer Treatment Trial II Group. Effect of Oral Voriconazole on Fungal Keratitis in the Mycotic Ulcer Treatment Trial II (MUTT II): A Randomized Clinical Trial. JAMA Ophthalmol. 2016 Dec 1;134(12):1365-1372. doi: 10.1001/jamaophthalmol.2016.4096. PMID 27787540
- [Derived] Prajna NV, Lalitha P, Rajaraman R, Krishnan T, Raghavan A, Srinivasan M, O'Brien KS, Zegans M, McLeod SD, Acharya NR, Keenan JD, Lietman TM, Rose-Nussbaumer J; Mycotic Ulcer Treatment Trial Group. Changing Azole Resistance: A Secondary Analysis of the MUTT I Randomized Clinical Trial. JAMA Ophthalmol. 2016 Jun 1;134(6):693-6. doi: 10.1001/jamaophthalmol.2016.0530. PMID 27054515
- [Derived] Rose-Nussbaumer J, Prajna NV, Krishnan T, Mascarenhas J, Rajaraman R, Srinivasan M, Raghavan A, Oldenburg CE, O'Brien KS, Ray KJ, Porco TC, McLeod SD, Acharya NR, Keenan JD, Lietman TM; Mycotic Ulcer Treatment Trial Group. Risk factors for low vision related functioning in the Mycotic Ulcer Treatment Trial: a randomised trial comparing natamycin with voriconazole. Br J Ophthalmol. 2016 Jul;100(7):929-932. doi: 10.1136/bjophthalmol-2015-306828. Epub 2015 Nov 3. PMID 26531051
- [Derived] Rose-Nussbaumer J, Prajna NV, Krishnan KT, Mascarenhas J, Rajaraman R, Srinivasan M, Raghavan A, Oldenburg CE, O'Brien KS, Ray KJ, McLeod SD, Porco TC, Lietman TM, Acharya NR, Keenan JD; Mycotic Ulcer Treatment Trial I Group. Vision-Related Quality-of-Life Outcomes in the Mycotic Ulcer Treatment Trial I: A Randomized Clinical Trial. JAMA Ophthalmol. 2015 Jun;133(6):642-6. doi: 10.1001/jamaophthalmol.2015.0319. PMID 25764482
- [Derived] Sun CQ, Prajna NV, Krishnan T, Mascarenhas J, Rajaraman R, Srinivasan M, Raghavan A, O'Brien KS, Ray KJ, McLeod SD, Porco TC, Acharya NR, Lietman TM. Expert prior elicitation and Bayesian analysis of the Mycotic Ulcer Treatment Trial I. Invest Ophthalmol Vis Sci. 2013 Jun 14;54(6):4167-73. doi: 10.1167/iovs.13-11716. PMID 23702779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 3, 2010, and December 31, 2011, patients were recruited from the Cornea Clinics at the Aravind Eye Care Hospitals in Madurai, Pondicherry, and Coimbatore in Tamil Nadu, India.
Period: Overall Study
Arm/Group | Topical Natamycin | Topical Voriconazole
Started | 162 | 161
3-week Visit | 155 (149 visited within pre-specified 3-week window (2.5-5 weeks); 6 had a second visit not within window) | 151 (144 visited within pre-specified 3-week window (2.5-5 weeks); 7 had a second visit not within window)
3-month Visit | 146 | 146
Completed | 141 | 143
Not Completed | 21 | 18
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 15 | 14
Not completed — Visit not within 3-month window | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Natamycin | Topical Voriconazole | Total
Number analyzed (Participants) | 162 | 161 | 323
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [39 to 58] | 45 [38 to 55] | 47 [39 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 67 | 140
  Male | 89 | 94 | 183
Region of Enrollment [Number; unit: participants]
  India | 162 | 161 | 323

OUTCOME MEASURES:

1. Primary Outcome: Best Spectacle-corrected logMAR Visual Acuity
Description: The primary analysis is best spectacle-corrected logMAR (logarithm of the Minimum Angle or Resolution) visual acuity, correcting for enrollment BSCVA and treatment arm in a multiple linear regression model. The pre-specified non-inferiority margin is less than 1.5 lines logMAR acuity. (Adjusted three-month visual acuity confidence bounds for the difference between the voriconazole and natamycin groups which meet or exceed 0.15 logMAR units would not permit noninferiority to be declared.) Note that this design also allows declaration of superiority (2-sided alpha of 0.05, corrected for an interim analysis).
Time Frame: 3 months from enrollment
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | Topical Natamycin | Topical Voriconazole
Number analyzed (Participants) | 141 | 143
logMAR | 0.39 [0.30 to 0.48] | 0.57 [0.48 to 0.65]
Statistical Analysis 1: Comparison: Topical Natamycin vs Topical Voriconazole; Test type: Non-Inferiority or Equivalence — The pre-specified non-inferiority margin is less than 1.5 lines logMAR acuity. (Adjusted three-month visual acuity confidence bounds for the difference between the voriconazole and natamycin groups which meet or exceed 0.15 logMAR units would not permit noninferiority to be declared.) Note that this design also allows declaration of superiority (2-sided alpha of 0.05, corrected for an interim analysis); p = 0.006, Regression, Linear; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.30 to -0.05]

2. Secondary Outcome: Best Spectacle-corrected logMAR Visual Acuity
Description: Best spectacle-corrected logMAR (logarithm of the Minimum Angle of Resolution) visual acuity at 3 weeks after enrollment, adjusting for enrollment BSCVA and treatment arm in a multiple linear regression model
Time Frame: 3 weeks after enrollment
Population: 306 total subjects (155 in natamycin arm, 151 in voriconazole arm) returned after enrollment for a second visit, but only 293 of those (149 in natamycin arm and 144 in voriconazole arm) visited within the 3-week window (2.5-5 weeks). Only those who visited within the window were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | Topical Natamycin | Topical Voriconazole
Number analyzed (Participants) | 149 | 144
logMAR | 0.49 [0.42 to 0.57] | 0.63 [0.56 to 0.70]

3. Secondary Outcome: Hard Contact Lens-corrected Visual Acuity Measured in logMAR
Description: Hard contact lens-corrected visual acuity measured in logMAR (logarithm of the Minimum Angle of Resolution) 3 months after enrollment
Time Frame: 3 months after enrollment
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | Topical Natamycin | Topical Voriconazole
Number analyzed (Participants) | 141 | 143
logMAR | 0.18 [0.11 to 0.26] | 0.30 [0.22 to 0.38]

4. Secondary Outcome: Size of Infiltrate/Scar
Description: Size of infiltrate/scar at 3 weeks and 3 months after enrollment, using enrollment infiltrate scar/size as a covariate
Time Frame: 3 weeks and 3 months after enrollment
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Topical Natamycin | Topical Voriconazole
Number analyzed (Participants) | 141 | 143
mm
  3 weeks from enrollment | 3.30 [3.15 to 3.48] | 3.44 [3.29 to 3.60]
  3 months from enrollment | 3.31 [3.15 to 3.48] | 3.52 [3.35 to 3.68]

5. Secondary Outcome: Time to Resolution of Epithelial Defect
Description: Time in days from enrollment to resolution of epithelial defect. For those subjects with more than 21 days to resolution, 21 days was used.
Time Frame: From enrollment to the time of resolution of epithelial defect
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Topical Natamycin | Topical Voriconazole
Number analyzed (Participants) | 162 | 161
days | 11.50 (7.60) | 11.50 (7.90)

6. Secondary Outcome: Minimum Inhibitory Concentration of Isolates
Description: Minimum inhibitory concentration (50th percentile) of fungal isolates to natamycin and voriconazole
Time Frame: 3 months after enrollment
Population: The population for analysis included only those subjects with positive fungal cultures and for whom Minimum Inhibitory Concentrations were available (108 subjects who were randomized to natamycin and 113 who were randomized to voriconazole).
Measure: Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | Topical Natamycin | Topical Voriconazole
Number analyzed (Participants) | 108 | 113
μg/ml | 4 [4 to 4] | 2 [1 to 2]

7. Secondary Outcome: Microbiological Cure at 6 Days
Description: Microbiological cure defined as no fungal growth on culture at 6 (+/-1) days from enrollment
Time Frame: 7 days after enrollment
Population: Of the 323 participants with smear-positive ulcers enrolled in the trial, 299 (92.6%) were scraped and cultured 6 days after enrollment - 155 in the natamycin arm, and 144 in the voriconazole arm.
Measure: Number; unit: participants
Arm/Group | Topical Natamycin | Topical Voriconazole
Number analyzed (Participants) | 155 | 144
participants | 23 | 69

ADVERSE EVENTS:
Arm/Group | Topical Natamycin | Topical Voriconazole
Serious Adverse Events (participants affected / at risk) | 42/162 | 82/161
Other Adverse Events (participants affected / at risk) | 10/162 | 27/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topical Natamycin (N=162) | Topical Voriconazole (N=161)
Corneal perforation (Eye disorders) | 10 | 15
Therapeutic penetrating keratoplasty (Eye disorders) | 13 | 29
Endophthalmitis (Eye disorders) | 0 | 2
Death (Eye disorders) | 1 | 1
Myocardial infarction or stroke (Cardiac disorders) | 0 | 1
Corneal perforation and/or TPK (Eye disorders) | 18 | 34
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topical Natamycin (N=162) | Topical Voriconazole (N=161)
Increase in hypopyon (>2mm) (Eye disorders) | 5 | 12
Increase in infiltrate size > 50% (Eye disorders) | 5 | 13
Progressive corneal thinning, <=50% of enrollment thickness (Eye disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No